CLINICAL TRIAL: NCT03907189
Title: Ambulation as a Factor on Oscillating Thermometry
Acronym: AFOOT
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Podimetrics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PCRT-0054P
Record Dates: First submitted 2019-03-26; First posted 2019-04-08 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Diabetic Neuropathy Peripheral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Emergent Inflammation: Subjects with emergent inflammation detected by Podimetrics RTM Mat within the last week.
- No Inflammation: Subjects with no emergent inflammation detected by Podimetrics RTM Mat within the last week.

SUMMARY:
This research study aims to better understand how the plantar temperature data collected by the Podimetrics RTM System corresponds to physical activity level in subjects.

DETAILED DESCRIPTION:
Subjects with prescription for monitoring with Podimetrics RTM System will be assigned activity monitors to track physical activity. Data from the Podimetrics RTM System and the activity monitor will be assessed after one month of use to determine any correlation between the two data sets and adherence to the use of activity monitor.

ELIGIBILITY:
Inclusion Criteria: Study subjects must

* Be at least 18 years old
* Not be pregnant
* Provide informed consent
* Have a prescription for monitoring with Podimetrics Remote Temperature Monitoring System

Exclusion Criteria:

* Be younger than 18 years old
* Unable to understand English
* Unable to provide consent
* At the discretion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study populations consists of patients at risk of diabetic foot ulcers and other inflammatory foot diseases with an existing prescription for monitoring with Podimetrics Remote Temperature Monitoring System.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-03-25 (Actual); Primary Completion 2020-12-10 (Estimated); Study Completion 2020-12-10 (Estimated)

PRIMARY OUTCOMES:
Correlation of foot temperature data and daily activity in patients with emergent inflammation. | 1 month
  The primary objective of the study is to examine whether temperature data from subjects with inflammation to the plantar foot as determined by the Podimetrics RTM System is correlated with activity as measured by the activity monitor.

SECONDARY OUTCOMES:
Correlation of foot temperature data and daily activity in patients without inflammation to the plantar foot. | 1 month
  The secondary objective of the study is to examine whether temperature data from patients without inflammation to the plantar foot as determined by the Podimetrics RTM System is correlated with subject activity as measure by the activity monitor.

OTHER OUTCOMES:
Usage rate for Podimetrics Mat | 1 month
  The objective is to record the number of distinct days on which subject uses Podimetrics Mat for thermometry reading.
Usage rate for the activity monitor | 1 month
  The objective is to record the percentage of time the subject uses the activity monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Petersen, MS,MBA, Principal Investigator — Podimetrics, Inc.
Locations (1):
- Podimetrics,Inc., Somerville, Massachusetts, United States